CLINICAL TRIAL: NCT02427828
Title: Continuous, Ambulatory, Non Invasive, Vital Sign Monitoring Using VRES of Cardiac Surgical Patients Following Discharge From Intensive Care. Impact on Detection of Physiological Deterioration
Brief Title: VRES Study in Two Phases to Monitor Cardiac Surgical Patients Following Discharge From ICU
Acronym: VRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OBS Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 011-0216-OTH
Record Dates: First submitted 2013-11-05; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): Assessment of Visensia Respiration Rate Estimation Service (product) to provide Respiration Rate from PPG signal, providing 3 vital signs (heart rate, oxygen saturation and respiration rate) to facilitate continuous Safety Index (VSI) calculation by Visensia, alongside standard routine intermittent observations (vital signs every 4 - 6 hours).
  Interventions: Device: Visensia Respiration Rate Estimation Service (VRES)
- Control Group (No Intervention): Using standard routine intermittent observation (vital signs every 4 - 6 hours) and calculation of NEWS/MEWS scores for early detection of patient deterioration.

INTERVENTIONS:
Device: Visensia Respiration Rate Estimation Service (VRES) — Medical device product to provide respiration rate from PPG signal
  Arms: Treatment Group

SUMMARY:
Failure to recognise deterioration early is a major cause of preventable deaths amongst hospital patients. The investigators wish to study whether continuous monitoring of 'vital signs' (pulse rate, breathing rate, and blood oxygen saturations) with computer modeled alerting to detect patient deteriorations can reduce cardiac arrest rate and critical care readmissions from the wards by alerting staff to clinical deteriorations more effectively than current paperbased systems.

Continuous monitoring of 'vital signs' can be achieved in two ways. Continuous monitoring of 'vital signs' has traditionally been restricted to the bedside because of the need for the patient to be connected by wires to the monitor.

More recently, advances in telemetry (wireless technology) have allowed the development of wearable devices which allow patients to mobilise freely, whilst constantly monitoring these 'vital signs'.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Papworth Hospital NHS Foundation Trust for routine cardiovascular surgery and who are discharged from ICU into the study ward (Mallard).

Exclusion Criteria:

* transplant surgery patients,
* VAD patients,
* children (less than 18 years old),
* prisoners (due to constant observation/security may bias normal level of care),
* patients who are subject to additional protections: this includes pregnant women, and persons with mental illness and learning disabilities,
* patients whose anatomy precludes the use of the required monitoring,
* patients who cannot understand written English (and where no translator is available),
* patients who are unable to give consent themselves,
* patients with learning difficulties who cannot understand the information to consent for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of ward cardiac arrests | Up to 72hours
  Duration of acute hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: John Mackay, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital, Papworth Everard, Cambridgeshire, United Kingdom